CLINICAL TRIAL: NCT01049659
Title: Effect of Iodine Supplementation and During Pregnancy on Neuropsychological Development of Children Assessed at 2 Years Old
Brief Title: Iodine Supplementation During Pregnancy and Neuropsychological Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09-PP-04
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Healthy; Iodine Deficiency; Pregnancy
Keywords: pregnancy; iodine deficiency; neuropsychological development
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- neuropsychological tests (Other): neuropsychological assessment of children around their second birthday
  Interventions: Behavioral: Neuropsychological test

INTERVENTIONS:
Behavioral: Neuropsychological test — Bayley test (version III) which provides several scales of development. Children are assessed just one time at two year old

SUMMARY:
The investigators have shown that Nice area, like most of France, remains an area of mild iodine deficiency. The investigators want to assess the potential benefit of early iodine supplementation during pregnancy in women with normal thyroid function on the neuropsychological development of their children assessed at the age of two with the Bayley test.

DETAILED DESCRIPTION:
Iodine is required for the synthesis of thyroid hormones. During pregnancy, iodine needs are increased to cover maternal and fetal thyroid hormones synthesis and the increased renal iodine clearance. Maternal hypothyroidism and/or severe iodine deficiency are associated to mental retardation in their offspring. Indeed, thyroid hormones and iodine are necessary for fetal brain development.

Iodine deficiency remains the first cause of preventable mental retardation. In France, preventive programs with salt iodine fortification are insufficient to eradicate iodine deficiency. In previous studies, we have shown that iodine deficiency is the rule for pregnant women in our area: 66 to 85% of women tested depending on the stage of pregnancy (Brucker-Davis 2004, Hieronimus et al 2009, abstract at the 2008 ETA and SFE meetings, article in preparation reporting results from our 2006 PHRC: Study of thyroid function during pregnancy with or without iodine supplementation).We will study the impact of early iodine supplementation in normal pregnant women on the neuropsychological development of their offspring assessed at 2 years of age. This is the follow-up of a cohort of children born to women enrolled in our 2006 PHRC. 110 healthy women have been included in this prospective study: they were seen early (median 8 weeks of gestation) and had strictly normal thyroid function tests, as well as no personal thyroid history. They were randomized into two groups: group A taking pregnancy vitamins without iodine supplementation (Oligobs GrossesseR 2 tablets/day) our group B taking the same vitamins but iodine fortified (Oligobs MaxiodeR 2 tablets per day, i.e. 150 mcg of iodine/day).

ELIGIBILITY:
Inclusion Criteria:

* children which mother were included in the precedent protocol(pregnancy vitamins with or without iodine)

Exclusion Criteria:

* children of more of 25 months old
* children with acute pathology
* children with chronic pathology

Ages: 23 Months to 25 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
neuropsychological test | one time mesure- just one visit in the study

CONTACTS AND LOCATIONS:
Overall Officials: Françoise BRUCKER-DAVIS, PhD, Principal Investigator — Nice University Hospital; Sylvie HIERONIMUS, PhD, Principal Investigator — Nice University Hospital
Locations (1):
- Endocrinology Department, Nice University Hospital, Nice, France